CLINICAL TRIAL: NCT00475462
Title: The Effectiveness of Metoprolol in the Prevention of Syncope Recurrence in Children and Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2004BA720A10
Record Dates: First submitted 2007-05-17; First posted 2007-05-21 (Estimated); Last update posted 2007-05-21 (Estimated); Status verified 2007-05

CONDITIONS: Syncope, Vasovagal
Keywords: Metoprolol and Syncope
MeSH Terms: conditions — Syncope, Vasovagal; Syncope | interventions — Metoprolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: metoprolol
Drug: conventional treatment

SUMMARY:
The purpose of this study to evaluate the effectiveness of metoprolol versus conventional treatment in the prevention of syncope recurrence in children and adolescents.

DETAILED DESCRIPTION:
Syncope is often a frustrating clinical problem seen in pediatric patients. Most pediatric syncope is benign, and vasovagal syncope (VVS) is the most common type of syncope seen in children . The diagnosis of VVS is established by history, often confirmed by tilt tests. A wide range of drugs has been proposed for VVS , with β-adrenergic blocking agents being first-line therapy. However, clinical studies have shown conflicting results in terms of therapy effectiveness. β-blockers have been claimed to be effective for 60% to 100% of young patients in many uncontrolled studies but not in most short- and long-term controlled studies . Sheldon et al., in a recent multicenter, double-blinded, placebo-controlled, randomized study of adult patients, reported that metoprolol was not effective in preventing VVS. To our knowledge, no pediatric randomized controlled trials with long-term follow-up have demonstrated the efficacy of β-blockers for the prevention of syncope.

ELIGIBILITY:
Inclusion Criteria:

* Children with a history of syncope were included if they had had at least three syncopal episodes per year and had a positive head-up tilt test result.

Exclusion Criteria:

* Patients were excluded if they had:

  * Other causes of syncope;
  * Cardiovascular and/or systemic disease;
  * Systolic blood pressure >130 mm Hg or diastolic blood pressure >90 mm Hg； or
  * History of asthma, impaired liver function, Ⅱ to Ⅲ degrees of atrioventricular block, sinus bradycardia < 40 beats/min, or other contraindications for β-blockers.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2001-07; Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
Our primary outcome variable was recurrence of syncope. | The primary endpoint was recurrence of syncope within 2 weeks after beginning therapy

CONTACTS AND LOCATIONS:
Overall Officials: Junbao DU, M.D., Study Director — Peking University First Hospital